CLINICAL TRIAL: NCT00310245
Title: Strategic Long Term, Immunologically Driven Treatment Interruptions in Patients on Effective HAART: a Controlled, Randomized Study
Brief Title: BASTA Study on STI in HIV Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG01
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2006-07-24 (Estimated); Status verified 2005-11

CONDITIONS: HIV Infection
Keywords: CD4-guided STI; Keywords:; HAART; Clinical outcome; Resistance; Costs; Prognostic factors; pulse therapy; treatment experienced; treatment interruption
MeSH Terms: conditions — HIV Infections | interventions — Treatment Interruption

INTERVENTIONS:
Procedure: STI (structured Treatment Interruption)

SUMMARY:
This is a single center, independent study. The primary objective is to compare efficacy and safety of continuing a conventional HAART in chronically infected HIV patients with a therapeutic strategy based on long term, immunologically driven treatment interruptions. Evaluation will be based on clinical, immunological and virological response.

Patients will be randomized in a ratio 1:2 to one of the two treatment arms:

Control group continuing the ongoing therapy STI group performing long term CD4 guided structured treatment interruptions In the STI arm patients will stay off therapy until their CD4 count will drop < 400 cells/mcL. At that time point patients will resume the HAART regimen they were assuming before STI and will continue HAART until they CD4 count will raise > 800 cells/mcL and their HIV-RNA will drop below the detection limit of 50 copies/ml. When both the CD4 count and the viral load will be within these pre-set values they will stop therapy again. There is no limit to the number of interruptions and re-start cycles during the study period The study is powered to evaluate equivalence between the two strategies under the assumption of a failure proportion in the control arm at each time point not greater than 5% and a maximum allowed difference of 15%.

DETAILED DESCRIPTION:
Study objectives

Primary objective of the study is:

To compare efficacy (clinical and immunological) and safety of continuing a conventional HAART in chronically infected HIV patients with a therapeutic strategy based on long term, immunologically driven treatment interruptions. To verify the risk of developing viral resistance

Secondary objectives are:

To verify the effect of the two strategies on metabolic parameters To verify the possibility to steadily discontinue antiretroviral therapy in patients that started it with baseline immunological values higher than those currently recommended by international guidelines for HIV treatment To identify predictive variables of the possibility to safely discontinue antiretroviral therapy To verify the dynamic of CD4 + loss and HIV replication after treatment interruption To verify costs connected to the strategy

Inclusion and exclusion criteria

a. Inclusion i. Age > 17 years ii. Informed consent signed iii. Effective ongoing treatment (HIV-RNA < 50 copies/ml). Treatment must be based on any triple drug therapy. Patients must be on the same steady therapy for at least 3 months.

iv. Current CD4 cell count above 800 cells/mcL b. Exclusion i. Childbearing or breastfeeding. Women of childbearing potential will be asked to adopt effective contraceptive methods or behaviors ii. Any ongoing grade 4 (WHO) AE or laboratory abnormality with the exclusion of cholesterol, triglycerides for which a grade 3 (AHA) level will be considered an exclusion criteria.

As the study wants to enroll patients strictly reflecting the population of HIV infected individuals, previous mono or dual therapies as well as the presence of co-morbidities such as HBV and HCV co-infection do not constitute exclusion criteria, but will be recorded

Study design

This is a randomized, controlled, open, comparative study. The trial will have a follow-up of 4 years.

Patients will be monitored according to the international and local guidelines for HIV infection as far as timing and type of laboratory and clinical controls. Laboratory exams will be decided locally and only a few key tests are required for the study. The timing of laboratory evaluation will be 1 and 2 months after each treatment interruption and thereafter every 2 months. All data will be stored in a computerized data-base.

Study arms and management of the study

Patients will be randomized in the ratio 1: 2 to one of the following treatment arms:

1. Continuing their ongoing HAART (control)
2. Long term treatment interruption (STI) Randomization will be accomplished locally according to a pre-determined, computer-generated random list.

In the control group, patients will be allowed to change therapy for virological, toxicological or personal reasons as well as to comply with new indications from international guidelines. All variation will be recorded. Patients changing therapy will be still included in the ITT analysis, but will be considered failures in the AT analysis. Patients stopping therapy, for any reason and not resuming it within 3 months will be considered as failures for both the AT analysis In the STI arm, patients will stay off therapy until their CD4 count drop < 400 cells/mcL (one measurement will be considered sufficient). At that time point patients will resume the HAART regimen they were assuming before the STI period (unless judged as no more of choice according to new international guidelines) and will continue HAART until their CD4 count raises > 800 cells/mcL and their plasma HIV-RNA drops below the detection limit of 50 copies/ml (one measurement will be considered sufficient). When both the CD4 count and the viral load will be within these pre-set values they will stop therapy again. There is no limit to the number of interruptions and re-start cycles during the study period 100 patients will be allocated in the STI arm and 30 patients in the control arm.

End points and evaluation criteria

The primary end-points for the evaluation of the main objective of the study can be divided in short term end points and long term end points:

The primary short term outcome measure will be the proportion of subjects maintaining at each time-point (every 4 months) a CD4 + cell count above 400 cells/mcL. The trial power is calculated on this end point.

On the long term, the primary outcome measure will be based on the occurrence of clinical end-points including: disease progression defined as the occurrence of any AIDS defining event and death. The occurrence of grade 4 (WHO) adverse events limiting the possibility to maintain the patient in the randomized arm will also be considered in AT analysis.

Virologic failure with the selection of resistance conferring mutations is the second long-term primary end-point. Genotypic tests will be performed in the case of HIV-RNA > 1000 copies/ml while on therapy for at least 6 months (in either group).

The secondary objectives of the study will be evaluated on the basis of:

Mean variation of blood cholesterol and triglycerides from baseline values. For these parameters the proportion of subjects with a value above grade 2 (AHA) will be also used as evaluation criteria.

Development of lipodystrophy or modification of a pre-existing lipodystrophy Time off therapy Economic evaluation Genotypic tests to be performed in the case of HIV-RNA > 1000 copies/ml while on therapy for at least 4 months or one month after each treatment interruption.

Duration of the study

Treatment will be continued for 4 years under the study conditions. Patients completing the study period and still responding to therapy will be kept on the same regimen.

Statistical evaluation of the study will be performed yearly.

Monitoring

Laboratory tests during the study period will be performed in he fasting state. The following tests and procedures are required and will be recorded in the electronic data base. It is also advised to perform on regular basis haemogram, renal function tests, blood glucose and amylase. Other test could be performed according to local needs or particular situations related to the specific management of single patients:

Baseline (all patients) i. Informed consent and treatment randomization ii. Biochemical analysis: ALT, AST, total cholesterol and HDL, triglycerides iii. CD4 count, CD8 count iv. Plasma HIV-RNA v. Clinical evaluation, anamnestic and demographic data: sex, age, risk factor for HIV infection, CDC AIDS classification, time on ART, time on current HAART, previous antiretroviral drugs, previous sub-optimal ARTs, current antiretroviral drugs, presence and grade of lipodystrophy, time with HIV-RNA below detection, nadir CD4, CD4 at start of antiretroviral therapy

1. month after each STI (only STI group) i. CD4 count, CD8 count, HIV-RNA
2. months after each STI (only STI group) i. Biochemical analysis: ALT, AST, cholesterol (total and HDL), triglycerides ii. CD4 count, CD8 count iii. Plasma HIV-RNA, Genotype iv. Clinical evaluation: disease progression, lipodystrophy assessment Every 2 months thereafter (STI group and control group) i. Biochemical analysis: ALT, AST, cholesterol (total and HDL), triglycerides ii. CD4 count, CD8 count iii. Plasma HIV-RNA iv. Clinical evaluation: disease progression, lipodystrophy assessment Additional tests

Additional tests will be requested in specific cases:

i. a second genotype after 4 months from the initiation of the STI period will be performed in all patients showing a major mutation in the genotype performed 2 months after STI start ii. a genotype will be performed in all patients either in the STI or in the control group showing a viral load above 1000 copies/ml after a continuous treatment period (on drugs) > 5 months.

Statistical considerations

The study is powered to evaluate equivalence between the two strategies under the assumption of a failure proportion in the control arm at each time point not greater than 5% and a maximum allowed difference of 15%. Equivalence will be defined on the basis of the 95% confidence interval.

According to this hypothesis with alfa = 5% and 1-beta = 80% a minimum of 70 patients will be needed. The primary analysis will be made according to the intention-to-treat approach and therefore no correction for eventual drop outs is needed.

In addition, a secondary per-protocol analysis will be performed. The primary outcome measure (the proportion of patients with CD4 + cell counts above 400 cells/mcL) will be analyzed by means of Chi-square or Fisher's exact test that will be used to analyze all other categorical variables, too. Time to treatment failure will be estimated using Kaplan-Meier product-limit estimates (that will be presented graphically). The log-rank test will be used to assess the difference between the survival curves for each arm, while ANOVA test and Student's t test will be used for continuous variables unless the variables will not be normally distributed, in which case the Mann-Whitney U tests will be used. Logistic regression analyses (forward stepwise model) will be used to evaluate the relationship between variables and outcome. Comparisons between pairs of groups will bee performed only in the case of a multiple test yielding a statistically significant result.

All tests will be two-sided and a P value inferior to 0.05 will be regarded as significant.

The analysis of data will be performed by the proposing Study Center with the SPSS statistical software package for Windows, version 10.0.

Drugs

This is a spontaneous study. It is proposed that all drugs will be dispensed according to standard procedures.

Data use

Data will be used for scientific purposes only. The analysis will be performed yearly. The type and timing of publication of data will be agreed among the participants to the study. The authorship of each presentation will be agreed among participants. All participants will be acknowledged as members of the study group.

ELIGIBILITY:
Inclusion Criteria:

i. Age > 17 years ii. Informed consent signed iii. Effective ongoing treatment (HIV-RNA < 50 copies/ml). Treatment must be based on any triple drug therapy. Patients must be on the same steady therapy for at least 3 months.

iv. Current CD4 cell count above 800 cells/L

Exclusion Criteria:

i. Childbearing or breastfeeding. Women of childbearing potential will be asked to adopt effective contraceptive methods or behaviors ii. Any ongoing grade 4 (WHO) AE or laboratory abnormality with the exclusion of cholesterol, triglycerides for which a grade 3 (AHA) level will be considered an exclusion criteria.

iii. Previous use of immunomodulatory agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2000-11; Study Completion 2005-11

PRIMARY OUTCOMES:
Proportion of subjects maintaining at each time-point a CD4 + cell count above 400 cells/mcL.
Occurrence of clinical end-points (AIDS defining event and death)
Virologic failure with the selection of resistance conferring mutations.

SECONDARY OUTCOMES:
Mean variation of blood cholesterol and triglycerides from baseline values. For these parameters the proportion of subjects with a value above grade 2 (AHA) will be also used as evaluation criteria.
Development of lipodystrophy or modification of a pre-existing lipodystrophy
Time off therapy
Economic evaluation
Genotypic tests to be performed in the case of HIV-RNA > 1000 copies/ml while on therapy for at least 4 months or one month after each treatment interruption.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Maggiolo, MD, Principal Investigator — Ospedali Riuniti, Bergamo
Locations (1):
- Antiviral Therapy Unit, Ospedali Riuniti, Bergamo, Bergamo, Italy

REFERENCES:
- [Result] Maggiolo F, Ripamonti D, Gregis G, Quinzan G, Callegaro A, Suter F. Effect of prolonged discontinuation of successful antiretroviral therapy on CD4 T cells: a controlled, prospective trial. AIDS. 2004 Feb 20;18(3):439-46. doi: 10.1097/00002030-200402200-00010. PMID 15090796